CLINICAL TRIAL: NCT05652595
Title: Double-blind, Randomized Comparative Cross-sectional Study of Pharmacodynamics and Pharmacokinetics of Drugs GP40141, Powder for Solution for Subcutaneous Administration, 250 µg (GEROPHARM LLC, Russia) and Enplate®, Powder for Solution for Subcutaneous Administration, 250 µg (Amgen Europe B.V. ., Netherlands) in Healthy Volunteers With a Single Subcutaneous Injection
Brief Title: Double-blind, Randomized Comparative Cross-sectional Study of Pharmacodynamics and Pharmacokinetics of Drugs GP40141
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GP40141-P4-31
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Pharmacodynamics; Pharmacokinetics; Bioequivalence
Keywords: romiplostim
MeSH Terms: interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, cross-over study of comparative pharmacodynamics and pharmacokinetics
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR Sequence (Experimental): first Intervention period - subjects are administered test medecine (GP40141) and in seconde Intervention period subjects are administered reference medecine (Nplate)
  Interventions: Drug: GP40141; Drug: Nplate
- RT Sequence (Experimental): first Intervention period subjects are administered reference medecine (Nplate) and in seconde Intervention period subjects are administered test medecine (GP40141)
  Interventions: Drug: GP40141; Drug: Nplate

INTERVENTIONS:
Drug: GP40141 — Once, at a dose of 3 mcg/kg, Subcutaneously in the shoulder area
  Other Names: romiplostim
Drug: Nplate — Once, at a dose of 3 mcg/kg, Subcutaneously in the shoulder area
  Other Names: romilostim

SUMMARY:
Bioequivalence Study of GP40141 (GEROPHARM) versus Enplate®. The study of comparative pharmacodynamics, pharmacokinetics and safety of drugs containing romiplostim in healthy volunteers after a single subcutaneous injection.

DETAILED DESCRIPTION:
The goal of this study, conducted as a double-blind, randomized, cross-over study of comparative pharmacodynamics and pharmacokinetics, is to compare pharmacodynamics, pharmacokinetics, and safety of drugs containing romiplostim - GP40141 and Nplate® in healthy volunteers after a single subcutaneous injection.

research objectives is:

1. Evaluate pharmacodynamic and pharmacokinetic parameters of active ingredients of preparations GP40141 and Enplate®.
2. Conduct a comparative analysis of pharmacodynamic and pharmacokinetic parameters of active substances drugs GP40141 and Enplate®.
3. Conduct a comparative analysis of data on adverse events (AE) and evaluate immunogenicity after a single subcutaneous administration of GP40141 versus Enplate®. A conclusion about the biosimilarity of drugs will be made by assessing 90% confidence intervals for the ratios of the geometric mean values of the primary pharmacodynamic parameters.

The safety of the compared drugs will be assessed by emergence and development of AE.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent form. Male aged 18 to 45 years. Verified diagnosis is "healthy" according to data Standard clinical, laboratory and Instrumental methods of examination.

The level of platelets count (according to the clinical blood test) at screening ranged from the lower threshold of reference values to 306×109/l (inclusive).

Body mass index between 18,5 and 30 kg/m2, with body weight 60-100 kg Consent to comply with an adequate method of effective contraception throughout the study.

The consent of volunteers to all restrictions imposed during the study. Russian Federation Citizens

Exclusion Criteria:

History of allergic problems/events. Hypersensitivity to heparin, romiplostim or any of the excipients of the drugs studied or E.coli protein.

Any acute and chronic diseases, including but not limited to cardiovascular system diseases, bronchopulmonary diseases, neuroendocrine systems diseases, as well as diseases of the gastrointestinal tract, liver, kidneys, blood.

Positive testing for hepatitis C (antibodies) or hepatitis B (surface antigen), HIV (antibodies to HIV-1/2), syphilis (antibodies to Treponema pallidum).

The WHO norms deviations of the heart rate (60-89), Sistolic BP (90-139 mm Hg), Diatolic BP (60-89 mm Hg), respiratory rate (12-20), body temperature (35.7 - 37.0 °C).

Abnormal ECG during screening. Abnormal results of laboratory methods research. Inaccessible veins of the upper extremities, vein thrombosis, thrombophlebitis in the anamnesis or in the family history of the next of kin, "compromised" veins due to frequent previous venipuncture.

Surgical interventions on the spleen, splenectomy in anamnesis. Acute infectious diseases in less than 4 weeks before the start of the study. Diseases of the blood, hematopoietic organs and disorders, involving the immune mechanism (ICD-10: D50-D89) in history.

History of arterial and venous thromboses. Presence of malignant (ICD-10: C00-C97) or unknown malignancy of neoplasms (ICD-10: D37-D48), as well as neoplasms in situ (ICD-10: D00-D09) within the last 5 years.

Regular intake of medications, including vitamins, herbal preparations, and dietary supplements, less than 2 weeks before the start of the study.

Incomplete recovery from surgery or surgery scheduled for the duration of the subject's participation in the study.

Significant loss of blood within 3 months prior to screening, including but not limited to blood donation or extended surgery or trauma resulting in the blood loss.

History of alcohol or drugs abuse or any indication of the regular use of more than 10 units of alcohol per week (1 Unit = 200 mL of wine or 500 mL of beer or 50 mL of alcohol 40%).

Positive test results for alcohol or drug use. Nicotine addiction, regular use of tobacco, including all types of electronic cigarettes, less than 6 months prior to screening.

Participation in a clinical trial of any drugs (including experimental) or experimental medical devices for 3 months or 5 half-lives, whichever is longer, before the study.

Dehydration due to diarrhea, vomiting, or other causes within the last 24 hours before the start of the study.

Any diet (for example, vegetarian, fasting, etc.) or lifestyle (including night work and extreme physical activity) that may interfere with the study.

Psychiatric disorders, history of epilepsy and seizures. Taking medications that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 30 days before the start of the study.

Volunteers who are obvious or likely, according to the investigator, are unable to understand and evaluate the information on this study as part of the process of signing informed consent, in particular regarding the expected risks and possible discomfort.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — males
Enrollment: 56 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
AUCplt | -45, -30, -15 min and days 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32 post injection
  the total area under the curve "amount platelets - time" in the time interval from "-45 minutes" to the moment t (day 32 after injection)
Pmax | -45, -30, -15 min and days 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32 post injection
  maximum number of platelets count (any time)

SECONDARY OUTCOMES:
Pmax/P0 | -45, -30, -15 min and days 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32 post injection
  ratio: maximum number of platelets count to the basal level of platelets
tPmax | -45, -30, -15 min and days 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32 post injection
  time to reach the maximum number of platelets count
AUC0-t | -15 min and 1, 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 hour post injection, and additionally 4, 5, 6, 8, 10, 12, 16, 20 days post injection
  total area under the curve "concentration of the active substance of the drug - time"
Cmax | -15 min and 1, 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 hour post injection, and additionally 4, 5, 6, 8, 10, 12, 16, 20 days post injection
  blood maximum concentration of the active substance of the drug
Tmax | -15 min and 1, 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 hour post injection, and additionally 4, 5, 6, 8, 10, 12, 16, 20 days post injection
  time to reach the maximum blood concentration (Cmax) of the active substance of the drug
T1/2 | -15 min and 1, 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 hour post injection, and additionally 4, 5, 6, 8, 10, 12, 16, 20 days post injection
  half-life of the active substance of the drug
AUC0-∞ | -15 min and 1, 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 hour post injection, and additionally 4, 5, 6, 8, 10, 12, 16, 20 days post injection
  total area under the curve "concentration of the active substance of the drug - time" time interval from -15 min to infinity, after the administration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Igor Mr Makarenko, PhD, Study Chair — GEROPHAM
Locations (1):
- Yaroslavl Region "Clinical Hospital No. 3", ,, Mayakovskogo st., 61, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makarenko I, Dorotenko A, Noskov S, Banko V, Saparova V, Khokhlov A, Zoreeva E, Nedorubov A, Zinnatulina B, Gefen M, Drai R. A randomized, double-blind, comparative study of the pharmacodynamics and pharmacokinetics of GP40141 (romiplostim biosimilar) and reference romiplostim in healthy male volunteers. Pharmacol Res Perspect. 2023 Oct;11(5):e01125. doi: 10.1002/prp2.1125. PMID 37740581